CLINICAL TRIAL: NCT01093820
Title: Documentation of Hemoglobin Kinetics in Response to Mircera® in Patients With Acute Myocardial Infarction (BEAT-STEMI Pilot)
Brief Title: Hemoglobin Kinetics in Response to Mircera® in Patients With Acute Myocardial Infarction
Acronym: BEATSTEMIPi
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010 DR 2029
Record Dates: First submitted 2010-03-16; First posted 2010-03-26 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: Acute Myocardial Infarction
Keywords: acute myocardial infarction; continuous erythropoetin receptor activator; Mircera; hemoglobin kinetics
MeSH Terms: interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epopoetinum beta (Experimental): Mircera® 150μg i.v., before / during reperfusion of the infarct related coronary artery followed by Mircera® 30μg s.c. at 1 and 2 months post-MI
  Interventions: Drug: methoxy-polyethyleneglycol epoetin beta

INTERVENTIONS:
Drug: methoxy-polyethyleneglycol epoetin beta — Mircera® 150μg i.v., before / during reperfusion of the infarct related coronary artery followed by Mircera® 30μg s.c. at 1 and 2 months post-MI
  Other Names: Mircera

SUMMARY:
Hypothesis:

Based on available pharmacokinetic data from healthy volunteers we hypothesize that the administration of a cumulative dose of 210μg of the continuous erythropoietin receptor activator, Mircera® (Roche), during 3 months post percutaneous coronary intervention (PCI) does not result in hemoglobin (Hb) levels >15 g/dl in patients with ST-segment elevation myocardial infarction (STEMI)

Design:

Prospective, open label single center pilot study

DETAILED DESCRIPTION:
This pilot trial will include 8 patients. The inclusion of 8 patients will allow to perform representative statistics of expected Hb kinetics in response to Mircera®.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age 18 - 80 years) with acute STEMI undergoing PCI

Main Exclusion Criteria:

* Hemoglobin levels >15g/dL
* history of a myeloproliferative syndrome
* thrombolysis for index infarction
* anticipated additional revascularization within 3 months
* cardiogenic shock

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients exceeding Hemoglobin (Hb) of 15 g/L within 3 months | three months
  measurement of Hb at baseline and month 1, 2 and 3

SECONDARY OUTCOMES:
Maximal change in Hb within 3 months relative to baseline | three months
  measurement of Hb at baseline and month 1, 2 and 3
Relative change in Hb from baseline to 1 months | first month
  measurement of Hb at baseline and month 1
Maximal change in Hematocrit (Hk) within 3 months relative to baseline | three months
  measurement of Hk at baseline and month 1, 2 and 3
change in platelet count within 3 months relative to baseline | three months
  measurement of platelet count at baseline and month 1, 2 and 3
Safety endpoints including all cause mortality,myocardial infarction,stroke,hospitalization,life threatening arrhythmias,thromboembolic events,stent thrombosis,poorly controlled hypertension despite therapy,seizures | three months
  follow-up at month 1, 2 and 3
Relative change in Hb from 1 to 2 months | second month
  measurement of Hb at month 1 and 2
Relative change in Hb from 2 to 3 months | third month
  measurement of Hb at month 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Pfisterer, Prof. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland